CLINICAL TRIAL: NCT07347080
Title: A Single-Center, Open-Label, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Exenatide Circular RNA-Lipid Nanoparticle Injection (CR059) in Chinese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Single-Center, Open-Label, Single Ascending Dose Study of Exenatide Circular RNA-Lipid Nanoparticle Injection (CR059) in Chinese Subjects With Type 2 Diabetes Mellitus
Acronym: CR059101
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Collaborators: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR059101
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: T2DM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exenatide Circular RNA-Lipid Nanoparticle Injection（CR059） (Experimental)
  Interventions: Drug: Exenatide Circular RNA-Lipid Nanoparticle Injection（ CR059））

INTERVENTIONS:
Drug: Exenatide Circular RNA-Lipid Nanoparticle Injection（ CR059）） — use one dose per person

SUMMARY:
Primary Objectives:

•To evaluate the safety and tolerability of a single dose of Exenatide Circular RNA-Lipid Nanoparticle Injection（CR059）in Chinese subjects with T2DM.

Secondary Objectives:

* To characterize the pharmacokinetic (PK) profile of a single dose of Exenatide Circular RNA-Lipid Nanoparticle Injection（CR059） in Chinese subjects with T2DM;
* To characterize the pharmacodynamic (PD) profile of a single dose of Exenatide Circular RNA-Lipid Nanoparticle Injection（ CR059） in Chinese subjects with T2DM;
* To evaluate the immunogenicity of a single dose of Exenatide Circular RNA-Lipid Nanoparticle Injection（ CR059） in Chinese subjects with T2DM;

Participants :

Diagnosed with T2DM for at least 3 months but less than 5 years, according to the Chinese Diabetes Society's diagnostic criteria

DETAILED DESCRIPTION:
This is a single-center, open-label, single ascending dose study designed to evaluate the safety, tolerability, PK, PD, and immunogenicity of Exenatide Circular RNA-Lipid Nanoparticle Injection（ CR059）in Chinese subjects with T2DM. It is planned to enroll 6-9 subjects.The study includes three dose cohorts (low, medium, high: 4 μg/kg, 8 μg/kg, 12 μg/kg). Each cohort plans to enroll 2-3 T2DM subjects. A single dose will be administered, with subjects observed in-hospital for at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female， 18≤age≤-65 years .
* Diagnosed with T2DM for at least 3 months but less than 5 years, according to the Chinese Diabetes Society's "Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes (2024 Edition)" diagnostic criteria.
* Patients who have failed treatment with diet and exercise alone, or metformin monotherapy, or a stable regimen for 12 weeks of metformin (dose ≥1500 mg/day or maximum tolerated dose ≥1000 mg/day) combined with one of the following oral antidiabetic drugs (or their fixed-dose combinations): sulfonylureas, glinides, alpha-glucosidase inhibitors, SGLT2 inhibitors, or thiazolidinediones (at ≥1/2 the maximum approved dose, or the recommended minimum maintenance dose for SGLT2 inhibitors e.g., empagliflozin 10mg, canagliflozin 100mg). Fasting Plasma Glucose (FPG) must be <13.0 mmol/L, and 7.5%≤HbA1c ≤ 10.0%.
* 18.5 kg/m²≤Body Mass Index (BMI) ≤40.0 kg/m² at screening and enrollment
* Subjects have no pregnancy plan from screening until 3 months after the last dose and are willing to use at least one effective method of contraception during the entire trial period until 3 months after the last dose.
* Able to understand and willing to sign the informed consent form, and fully understand the trial content, procedures, and potential adverse reactions.
* Able to complete the trial according to the protocol requirements.

Exclusion Criteria:

* Diagnosis of type 1 diabetes, diabetes due to pancreatic injury, or specific types of diabetes due to other diseases (e.g., acromegaly or Cushing's syndrome).
* History of acute diabetic complications, such as ketoacidosis or hyperosmolar coma, within 6 months before screening.
* Presence of severe chronic diabetic complications (e.g., proliferative diabetic retinopathy, severe diabetic neuropathy, diabetic foot, etc.) within 6 months before screening, deemed by the investigator as unsuitable for participation.
* Allergic constitution (allergy to ≥2 types of drugs or foods) or keloid tendency, or clear history of drug allergy, or investigator suspects potential allergy to the investigational product or its components or similar drugs.
* Fasting plasma glucose <3.9 mmol/L at screening or before enrollment, and/or history of ≥2 episodes of severe hypoglycemia or recurrent symptomatic hypoglycemia within 6 months before screening.
* History or presence of Cushing's syndrome, polycystic ovary syndrome, or other hereditary endocrine diseases, or obesity secondary to factors such as hormones.
* Use of weight-control medications or weight-loss surgery within 3 months before screening, or weight fluctuation exceeding 5% within 3 months.
* Clinically significant abnormal TSH, FT3, or FT4 at screening, or previous diagnosis of thyroid dysfunction, deemed unsuitable by the investigator.
* Personal or family history of multiple endocrine neoplasia type 2; personal or family history of medullary thyroid carcinoma; or thyroid nodules classified as C-TIRADS category 4 or higher on ultrasound.
* History or presence of malignant tumors (except cured basal cell carcinoma or cervical carcinoma in situ).
* History of thrombotic diseases (e.g., deep vein thrombosis, pulmonary embolism, stroke), known bleeding diathesis or coagulation dysfunction, major thrombotic event within 6 months, or any coagulation parameter ≥1.5x ULN, or clinically significant abnormal coagulation function deemed unsuitable by the investigator.
* Long-term use (over 1 month) or current use of anticoagulants (e.g., warfarin, rivaroxaban, dabigatran) or antiplatelet drugs (e.g., aspirin, clopidogrel) before screening.
* Diagnosis of significant cardiovascular or cerebrovascular disease within 6 months before screening, including but not limited to acute stroke, transient ischemic attack (TIA), acute coronary syndrome, coronary heart disease, heart failure, arrhythmia requiring treatment, etc.
* History of gout or gout attack within 6 months before screening or before enrollment.
* Untreated or poorly controlled hypertension (systolic BP >160 mmHg and/or diastolic BP >100 mmHg) at screening or before enrollment. Patients on antihypertensive therapy must have a stable regimen and dose for 1 month. If BP criteria are not met at screening/enrollment, one re-test is allowed. Exclusion if both readings fail.
* Heart rate at rest (after at least 10 min) <50 bpm or >100 bpm at screening or before enrollment. One re-test is allowed. Exclusion if both readings fail.
* PR interval >210 ms and/or QRS complex duration >120 ms, and/or QTcF >450 ms at rest at screening or before enrollment. If criteria not met, repeat ECG twice on the same day; use the average of 3 measurements for judgment.
* History of clinically significant chronic or acute exacerbating respiratory diseases, including but not limited to asthma, COPD (excluding obstructive sleep apnea).
* History of severe gastrointestinal disease (e.g., active ulcer, gastroparesis, pyloric obstruction, inflammatory bowel disease) within 6 months before screening or before enrollment, or gastrointestinal surgery, or long-term use of drugs directly affecting GI motility due to chronic GI disease, deemed unsuitable by the investigator.
* Severe renal disease or estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73m² (CKD-EPI formula) at screening or before enrollment.
* Serum amylase or lipase >3x Upper Limit of Normal (ULN) at screening or before enrollment, or history/known chronic pancreatitis, acute pancreatitis, pancreatic injury.
* History of cholelithiasis, acute or chronic cholecystitis (except those with no residual biliary stones post-treatment or post-cholecystectomy without sequelae, deemed eligible by the investigator).
* Severe dyslipidemia, with LDL-C ≥4.40 mmol/L or triglycerides (TG) ≥5.65 mmol/L at screening or before enrollment. If on lipid-lowering therapy, regimen and dose must be stable for 1 month.
* Clear history of psychiatric disorders (e.g., depression, schizophrenia, bipolar disorder) within 2 years before screening.
* Major surgery within 1 month before screening, or presence of severe infection or active inflammation.
* History of blood donation >400 mL, transfusion, or blood loss within 90 days before screening or before enrollment.
* Any of the following laboratory abnormalities at screening or before enrollment: 1. ALT or AST >2x ULN; 2. Total Bilirubin >1.5x ULN; 3. Calcitonin ≥35 pg/mL; 4. Hemoglobin <110 g/L (female) or <120 g/L (male); 5. Clinically significant abnormal platelet count; 6. Clinically significant abnormal white blood cell or neutrophil count;
* Use of any approved or unapproved weight-affecting drugs or products within 3 months before screening, including but not limited to orlistat, phentermine-topiramate, naltrexone-bupropion, systemic corticosteroids, antidepressants (SSRIs, SNRIs, tricyclics, tetracyclics), antipsychotics/sedatives (e.g., imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid, lithium), etc.
* Use of any DPP-4 inhibitor, or GLP-1, GIP, GCG receptor agonists, or FGF-21 within 6 months before screening.
* History of bariatric surgery (except liposuction/abdominoplasty >1 year prior).
* Participation in any drug or medical device clinical trial within 3 months before screening or before enrollment (except screen failures).
* Positive serology for HBsAg, anti-HCV antibody, anti-TP antibody, or anti-HIV antibody at screening.
* History of drug abuse and/or alcoholism (weekly alcohol intake >14 units) within 6 months before screening
* Positive urine drug screen or alcohol breath test at screening.
* Pregnant or lactating females, or subjects using oral contraceptives.
* Intolerance to venipuncture or history of needle syncope, blood-injury syncope.
* Any other physiological, psychological, or situational condition deemed by the investigator as unsuitable for trial participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the first dosing (Day 1 ) of study drug until completion of the post treatment follow-up visit(Day 36)
  Adverse events (AEs) / Serious adverse events (SAEs) will be collected via:
  Laboratory tests (including complete blood count, blood biochemistry, glucagon, lipase, amylase, urinalysis, coagulation function, high-sensitivity C-reactive protein, inflammatory factors); Vital signs (blood pressure, pulse rate, body temperature, respiration); Physical examinations (including skin, mucous membranes, lymph nodes, head and neck, chest, abdomen, spine and extremities, and musculoskeletal tissues); 12-lead electrocardiogram (12-lead ECG, including PR interval, QRS duration, QTcF interval); Abnormalities observed by the investigator; Subject-reported complaints.

SECONDARY OUTCOMES:
Pharmacokinetic | From the first dose (Day 1 ) of study drug until Day 36
  Cmax
Pharmacokinetic | From the first dose (Day 1 ) of study drug until Day 36
  Tmax
Pharmacokinetic | From the first dose (Day 1 ) of study drug until Day 36
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration（AUC0-last）
Pharmacokinetic | From the first dose (Day 1 ) of study drug until Day 36
  Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC0-inf)
Pharmacokinetic | From the first dose (Day 1 ) of study drug until Day 36
  Apparent Clearance (CL/F)
Pharmacokinetic | From the first dose (Day 1 ) of study drug until Day 36
  Apparent Volume of Distribution (VZ/F)
Pharmacokinetic | From the first dose (Day 1 ) of study drug until Day 36
  Elimination Half-Life (t1/2)
Anti-Drug Antibodies | Day 1 (first dosing day)、Day 15、Day 29
  ADA positivity rate
Pharmacodynamics | From the baseline(Day 2)until completion of the post treatment follow-up visit (Day 36)(Day 1 :first dosing day)
  Plasma Glucose
Pharmacodynamics | From the baseline(Day 2)until completion of the post treatment follow-up visit(Day 36)(Day 1 :first dosing day)
  Serum C-peptide
Pharmacodynamics | From the baseline(Day 2)until completion of the post treatment follow-up visit(Day 36)(Day 1 :first dosing day)
  Serum insulin
Anti-Drug Antibodies | Day 1(first dosing day)、Day 15、Day 29
  ADA titer

IPD SHARING:
Plan to Share IPD: Yes
underlie the results reported in this study-including demographics, baseline characteristics, efficacy, and safety data-will be shared with researchers who provide a methodologically sound proposal, starting 6 months after publication of the primary outcomes in a peer-reviewed journal.
Supporting Information: Analytic Code
Time Frame: Starting 6 months after publication of the primary outcomes in a peer-reviewed journal.The data will remain available for access for a period of 24 months.
Access Criteria: Access is restricted to academic researchers for non-commercial, scientific purposes
URL: https://register.clinicaltrials.gov/prs/beta/studies/S000GLP800000027/protocol/ipdSharing?edit=true